CLINICAL TRIAL: NCT05057871
Title: Efficacy of Pulse Electromagnetic Field Therapy (PEMF) in Patients With Subacromial Impingement Syndrome: A Randomized Study of Double Blınd With Sham Control
Brief Title: Efficacy of Pulse Electromagnetic Field Therapy (PEMF) in Patients With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Oğuzhan Kandemir, Research Assistant Doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUBIMPPEMF2021
Record Dates: First submitted 2021-09-17; First posted 2021-09-27 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Shoulder Pain; Musculoskeletal Diseases; Subacromial Impingement Syndrome; Shoulder Injuries and Disorders
Keywords: Pulse Electromagnetic Field Therapy; Subacromial Impingement Syndrome; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain; Musculoskeletal Diseases; Shoulder Impingement Syndrome; Shoulder Injuries; Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEMF+exercise (Experimental): A total of 20 sessions of pulse electromagnetic field therapy using an electromagnetic field device (ASA Pmt Quatro Pro, ASA Srl Via A.Volta 9-36057, Italia), five times a week and once a day for four weeks, were applied to the patients. The patients were then given a daily exercise program once a day by a physiotherapist.
  Interventions: Device: Pulse electromagnetic field therapy
- Sham PEMF+exercise (Sham Comparator): Sham therapy was applied in five sessions a week for four weeks, with a total of 20 sessions, with no current flowing through the device. This was followed by the exercise programs described above, performed once a day with the physiotherapist.
  Interventions: Device: Sham pulse electromagnetic field therapy

INTERVENTIONS:
Device: Pulse electromagnetic field therapy — It was applied with an electromagnetic field device (ASA Pmt Quatro Pro, ASA Srl Via A.Volta 9-36057 Italia) at 50 Hz frequency, 85 Gauss (8.5 milliTesla) intensity and for 30 minutes. The treatment period was 5 days a week for 4 weeks, in total. It was applied as 20 sessions.
  Therapeutic Exercise As a therapeutic exercise program; active shoulder ROM, isometric and progressive strengthening exercises for shoulder girdle muscles, codman pendulum exercises will be performed. It was planned to implement a total of 20 sessions 5 days a week for 4 weeks, for approximately 30 minutes. Exercises will be performed by a trained (at least 5 years experienced) physiotherapist, three times a day, in 3 sets, 10 repetitions.
  Arms: PEMF+exercise
Device: Sham pulse electromagnetic field therapy — Sham pulse electromagnetic field therapy was applied five sessions a week for four weeks, for a total of 20 sessions a day, using electromagnetic field device (ASA Pmt Quatro Pro, ASA Srl Via A.Volta 9-36057 Italy) without current flowing through the device.
  Therapeutic Exercise As a therapeutic exercise program; active shoulder ROM, isometric and progressive strengthening exercises for shoulder girdle muscles, codman pendulum exercises will be performed. It was planned to implement a total of 20 sessions 5 days a week for 4 weeks, for approximately 30 minutes. Exercises will be performed by a trained (at least 5 years experienced) physiotherapist, three times a day, in 3 sets, 10 repetitions.
  Arms: Sham PEMF+exercise

SUMMARY:
The aim of our study is to investigate the effectiveness of Pulse Electromagnetic Field Therapy (PEMT) versus placebo on pain, quality of life, shoulder function and isokinetic assessment, and muscle strength in the treatment of subacromial impingement syndrome.

DETAILED DESCRIPTION:
Shoulder pain is one of the common health problems. It ranks third among musculoskeletal problems after low back and neck pain. Subacromial Impingement Syndrome (SIS) is the most common cause of shoulder pain. SIS is a pathology resulting from mechanical repetitive compression and inflammation of the supraspinatus tendon, subacromial-subdeltoid bursa, and biceps tendon located under the acromion and coracoacromial ligament. SIS is characterized by functional limitation of the shoulder with gradual limitation of both active and passive glenohumeral movement due to compression of the subacromial structures. Pain in the anterior shoulder region, which is exacerbated by elevation of the shoulder joint or overhead activities, and limitation of range of motion are the main reasons for the decrease in quality of life in patients with SIS.

The most common symptom of SIS is pain. The pain is usually at night and radiates to the anterior aspect of the shoulder. Night pain often occurs when lying on the affected side and is typically in the deltoid region. Symptoms usually increase with abduction, elevation, or overhead activities. Patients often complain that they have difficulty reaching their back while dressing. Active movements may be restricted due to pain.

Analgesics and nonsteroidal anti-inflammatory drugs (NSAIDs), steroid injections, physical therapy methods, exercise and surgical procedures are used in the treatment of shoulder pain. Superficial hot and cold applications, analgesic currents, ultrasound, extracorporeal shock wave therapy (ESWT), magnetotherapy, laser and acupuncture are preferred as treatment options.

Magnetotherapy is a treatment method based on magnetic field interaction. As a result of pulsed or alternating electromagnetic fields, an electrical current occurs in the tissues. Pulse magnetotherapy has three physical mechanisms known to be effective in living tissue: Magnetic induction, magneto-mechanical effects, and electronic interactions. Effects of magnetic field application are vasodilation, analgesic effect, anti-inflammatory effect, acceleration of healing, antiedematous effect. Magnetotherapy increases the oxygen release of erythrocytes and provides oxygenation of the tissues. This causes a decrease in toxins in the damaged area, an increase in vital nutrients and endorphins. With this physiological change, magnetic energy decreases the pain receptor sensitivity that sends a message to the brain. With this treatment method, pain reduction is achieved, while joint mobility increases.

This study was designed as a double-blind, prospective, placebo-controlled, randomized study. Participants were randomized into 2 groups: PEMF + therapeutic exercise, sham PEMF + therapeutic exercise.

Shoulder range of motion, Visual Pain Scale (VAS), SF (Short form) -36 Quality of Life Scale, Constant Murley Scale, Shoulder pain and disability index, upper extremity muscle strength measurement with Isomed 2000 isokinetic device) will be evaluated. It was planned that the evaluations were made and recorded by a blinded physician to the groups at the beginning of the treatment, at the end of the treatment and at the 3rd month controls.

ELIGIBILITY:
Inclusion Criteria:

1. Shoulder pain for at least 6 weeks in the 30-65 age range
2. Positivity of shoulder impingement tests on examination(Neer test, Hawkins Kennedy test)
3. Findings related to subacromial impingement syndrome in MRI

Exclusion Criteria:

1. Pregnancy
2. Inflammatory rheumatologic diseases
3. Malignity
4. Having received physical therapy and rehabilitation for the shoulder area in the last 3 months
5. Local injection therapy to the shoulder area in the last 6 months
6. History of trauma, history of surgery, history of fracture in the aching shoulder region in the last 6 months
7. Adhesive capsulitis, calcification findings in the rotator cuff tendons exceeding 2 cm, findings of full-thickness total rotator cuff rupture in magnetic resonance (MR) imaging, presence of osteoarthritis findings and labral pathologies in imaging of the acromioclavicular joint or glenohumeral joint, presence of benign malignant lesions
8. cervical radiculopathy
9. Cervical myofascial pain syndrome
10. cardiac pacemaker
11. bleeding diathesis
12. Body implant with electronic or battery system
13. Acute infections
14. tuberculosis

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline visual analog scale (VAS) shoulder pain rest movement at 4th and 12th week | up to 12th week
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.

SECONDARY OUTCOMES:
Change from baseline quality of life (short form 36 (SF-36)) at 4th and 12th weeks | up to 12th week
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Total score was between 0 ( disability) and 100 (no disability). Every subgroup of the questionnaire has a score scale between 0 and 100. Every increase in the subgroup of SF-36 questionnaire, which is a positive scoring system, indicates increase in quality of life related to health.
range of motion | up to 12th week
  In shoulder range of motion measurement, flexion and abduction will be recorded, including active and passive measurements of the shoulder with a goniometer.Shoulder internal and external rotation measurements will be recorded while the patient's shoulder is abducted at 90 degrees and the elbow is flexed at 90 degrees.
Change from baseline Constant Murley Score (C-MS) at 4th and 12th weeks | up to 12th week
  The Constant-Murley Shoulder Score (C-M Score) is a clinical and functional assessment scale that evaluates the functional status of a normal, diseased or treated shoulder. Comparisons can be made in pre-treatment and post-treatment follow-up. Evaluated parameters were pain (15 points), activities of daily living (20 points), ROM (40 points), and strength (25 points).Scoring that measures the functionality of the shoulder consists of 100 points in total. C-M score; It is classified as excellent (90-100), good (80-89), moderate (70-79) and poor (<70).
Change from baseline Shoulder Pain and Disability Index(SPADI) at 4th and 12th weeks | up to 12th week
  It is a two-part scale that evaluates pain and function.The first part questions pain, the second part questions disability. In the pain section consisting of 5 items, the pain felt during activities of daily living is measured using a 10-unit VAS, and in the disability section, the difficulty encountered during activities of daily living is measured in the 8-item disability section. The score of both sections and the total score are calculated with a special formula.
Change from baseline upper extremity muscle strength with isokinetic device at 4th and 12th weeks | up to 12th week
  Isokinetic contraction; It is defined as contraction at a constant rate throughout the entire range of motion and at an equal rate at all angles of motion. No matter how hard a person moves the device, they can never exceed the predetermined speed (for example, 90 degrees per second). It is advantageous that the desired muscle or muscle groups can be evaluated in isolation and that the measurements are comparable. The isokinetic strength assessment of the patients during internal and external rotation of the shoulder will be made with an isokinetic device (IsoMed 2000, isokinetic dynamometer, Germany). Measurements will be made by a physiotherapist with at least 5 years of device experience. Measurements will be made in 10 repetitions to increase reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda MD ADAR, Principal Investigator — Afyonkarahisar Health Sciences University; Oğuzhan MD KANDEMİR, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michener LA, Walsworth MK, Burnet EN. Effectiveness of rehabilitation for patients with subacromial impingement syndrome: a systematic review. J Hand Ther. 2004 Apr-Jun;17(2):152-64. doi: 10.1197/j.jht.2004.02.004. PMID 15162102
- [Background] Galace de Freitas D, Marcondes FB, Monteiro RL, Rosa SG, Maria de Moraes Barros Fucs P, Fukuda TY. Pulsed electromagnetic field and exercises in patients with shoulder impingement syndrome: a randomized, double-blind, placebo-controlled clinical trial. Arch Phys Med Rehabil. 2014 Feb;95(2):345-52. doi: 10.1016/j.apmr.2013.09.022. Epub 2013 Oct 15. PMID 24139986
- [Background] Guo L, Kubat NJ, Isenberg RA. Pulsed radio frequency energy (PRFE) use in human medical applications. Electromagn Biol Med. 2011 Mar;30(1):21-45. doi: 10.3109/15368378.2011.566775. PMID 21554100
- [Background] Pribicevic M, Pollard H, Bonello R, de Luca K. A systematic review of manipulative therapy for the treatment of shoulder pain. J Manipulative Physiol Ther. 2010 Nov-Dec;33(9):679-89. doi: 10.1016/j.jmpt.2010.08.019. Epub 2010 Oct 18. PMID 21109059
- [Derived] Kandemir O, Adar S, Dundar U, Toktas H, Yesil H, Eroglu S, Eyvaz N. Effectiveness of Pulse Electromagnetic Field Therapy in Patients With Subacromial Impingement Syndrome: A Double-Blind Randomized Sham Controlled Study. Arch Phys Med Rehabil. 2024 Feb;105(2):199-207. doi: 10.1016/j.apmr.2023.09.020. Epub 2023 Oct 31. PMID 37820844